CLINICAL TRIAL: NCT01704781
Title: A Double-blind Placebo Controlled Immunogenicity Study of Vacc-4x + Lenalidomide Versus Vacc-4x With an Initial Open-label Dose Escalation Assessment of Lenalidomide in HIV-1-infected Subjects on Antiretroviral Therapy (ART).
Brief Title: Vacc-4x + Lenalidomide vs. Vacc-4x +Placebo in HIV-1-infected Subjects on Antiretroviral Therapy (ART)
Acronym: IMID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bionor Immuno AS (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CT-BI Vacc-4x/IMiD-2010/1
Record Dates: First submitted 2012-09-11; First posted 2012-10-11 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2014-10

CONDITIONS: HIV-1 Infection
Keywords: CD4; Clinical trial; Dose escalation assessment lenalidomide; Human immunodeficiency virus-1 (HIV-1); HIV; Immunomodulatory; Infection; Lenalidomide; Phase I/II; Vaccine; Vacc-4x
MeSH Terms: conditions — Infections | interventions — Lenalidomide; Vacc-4x; sargramostim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part A: lenalidomide dose escalation (Experimental): All patient receive intradermal Vacc-4x (1.2 mg) given with Leukine® (rhu-GM-CSF) (0.06 mg) and oral lenalidomide in a dose escalation (3+3) design.
  Dose level -1: 2.5 mg Lenalidomide (CC-5013) in the event Dose level 1 is non tolerated dose (NTD) Dose level 1(start): 5 mg Lenalidomide (CC-5013) Dose level 2: 10 mg Lenalidomide (CC-5013) Dose level 3: 25 mg Lenalidomide (CC-5013)
  Interventions: Drug: Lenalidomide; Drug: Vacc-4X; Drug: rhuGM-CSF
- Part B: lenalidomide (Experimental): Intradermal Vacc-4x (1.2 mg) given with Leukine® (rhu-GM-CSF) (0.06 mg) and oral lenalidomide for 6 immunizations (visit 2, 3, 4, 5, 6 and 7) & lenalidomide (dose determined in Part A) two days prior to and at the day of immunization.
  Interventions: Drug: Lenalidomide; Drug: Vacc-4X; Drug: rhuGM-CSF
- Part B: lenalidomide placebo (Placebo Comparator): Intradermal Vacc-4x (1.2 mg) given with Leukine® (rhu-GM-CSF) (0.06 mg) and oral lenalidomide for 6 immunizations (visit 2, 3, 4, 5, 6 and 7) & lenalidomide placebo two days prior to and at the day of immunization.
  Interventions: Drug: Lenalidomide placebo; Drug: Vacc-4X; Drug: rhuGM-CSF

INTERVENTIONS:
Drug: Lenalidomide — In Part A a dose escalation design is used (2,5; 5; 10; 25 mg). Part B will use the dose confirmed by Part A
  Other Names: Lenalidomide capsule
  Arms: Part A: lenalidomide dose escalation; Part B: lenalidomide
Drug: Lenalidomide placebo — Capsules are identical to the active Lenalidomide capsules used.
  Other Names: placebo
  Arms: Part B: lenalidomide placebo
Drug: Vacc-4X — Vacc-4x is a peptide-based HIV immunotherapy administered intradermally. Vacc-4x peptides are reconstituted in sterile water.
  Other Names: Combination of Vacc-10, Vacc-11, Vacc-12 and Vacc-13.
Drug: rhuGM-CSF — Granulocyte macrophage colony stimulating factor as a local adjuvant
  Other Names: Leukine®

SUMMARY:
During the course of HIV infection the number of CD4 cells decreases, resulting in a reduced immunological response and ultimately immune deficiency. Vacc-4x is a peptide-based HIV immunotherapy and the primary objective is to strengthen the immune system's response to HIV p24. By adding Lenalidomide, an immunomodulatory agent, as a supporting drug, it is anticipated that the effect of Vacc-4x might be enhanced.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV) infects the CD4 subset of T-cells that are critical for initiating immune responses to infection. The level of CD4 cells in the blood is a marker of a patient's immunological status. The number of CD4 cells decreases in the course of the HIV infection and results in a reduced immunological response and eventually immune deficiency.

Vacc-4x is one of the few peptide-based therapeutic vaccines tested, and consists of four, slightly modified HIV Gag p24 consensus peptides. Vacc-4x was first tested by intradermal injections using GM-CSF as adjuvant. A recent multinational placebo-controlled study found improvement of vaccine-specific T cell immunity and decrease in viral loads (presented at the AIDS vaccine 2011 conference, Bangkok).

Lenalidomide (CC-5013) is a substance in the class of immunomodulatory agents. The lenalidomide mechanism of action includes anti-neoplastic, pro-erythropoietic, and immunomodulatory properties. Lenalidomide inhibits proliferation of certain hematopoietic tumor cells, enhances T cell- and Natural Killer (NK) cell-mediated immunity and increases the number of NK T cells.

The anti-HIV p24 immune response resulting from Vacc-4x immunization could in combination with ART potentially improve immune reconstitution in patients who have not fully regained a healthy CD4 level (> 600 x106/L). Adding the immunomodulatory agent Lenalidomide (CC-5013) to Vacc-4x immunization could enhance the immune response to Vacc-4x and further strengthen immune reconstitution.

ELIGIBILITY:
Inclusion Criteria:

1. Men, age ≥ 18 and ≤ 55 years at the time of screening.
2. Women, age ≥ 50 and ≤ 55 years at the time of screening, who are not of childbearing potential (see Exclusion criteria, point 9). Childbearing status must be documented.
3. Clinically stable on ART for the last 18 months (changes in therapy are allowed as long as the viral load is stable).
4. Well controlled with no treatment failure due to ART resistance in the past
5. Screening plasma viral load (HIV-1 RNA) less than 50 copies/mL for the last six months. If screening value is between 50-500 copies/mL rescreening is allowed. Single blips (up to 500 copies/mL) are allowed.
6. Screening CD4 cell count ≥ 200x10^6 cells/L and ≤500x10^6 cells/L. (Rescreening is allowed)
7. Laboratory test results within these ranges: Absolute neutrophil count (ANC) >1.0x10^9 /L, Platelet count >75x10^9 /L and eGRF (MDRD) >60 mL/min
8. Signed informed consent
9. Willingness to adhere to Global Pregnancy Prevention Risk Management Plan Lenalidomide

Exclusion Criteria:

1. Reported pre-study AIDS-defining illness within the previous year
2. Malignant disease.
3. On chronic treatment with immunosuppressive therapy.
4. Autoimmune disorders, present or in the past if there is an increased risk of disease exacerbation.
5. Unacceptable values of the hematologic and clinical chemistry parameters (including those associated with hemophilia), as judged by the Investigator or the Sponsor (or designee), including creatinine values >1.5x upper limit of normal (ULN), and AST (SGOT), ALT (SGPT), and alkaline phosphatase values >2.5x ULN.
6. Concurrent chronic active infection such as viral hepatitis B or C or tuberculosis.
7. Previous thromboembolic events or patient is currently immobilized
8. Sexually active subjects who do not adhere to Global Pregnancy Prevention Risk Management Plan Lenalidomide
9. Current participation in other clinical therapeutic studies.
10. Females of childbearing potential will be excluded from this trial. A female of childbearing potential (FCBP) is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e. has had menses at any time in the preceding 24 consecutive months).
11. The development of erythema nodosum if characterized by a desquamating rash while previously
12. Incapability of compliance to the treatment protocol, in the opinion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Krogsgaard, Study Director — Bionor Pharma ASA, Kronprinsesse Märthas Plass 1, P.O. Box 1477 Vika, NO-0116 Oslo, Norway
Locations (4):
- Germany (4):
  - University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg
  - EIPMED - Gesellschaft fűr epidemiologische und klinische Forschung in der Medizin mbH Rubensstrasse 125, Berlin, State of Berlin
  - Charite Campus, Virchow-Klinikum Medizinische Klinik mit Schwerpunkt Infektiologie Station 59 (Suedring 11) Augustenburger Platz 1, Berlin, State of Berlin
  - Klinik I für Innere Medizin Klinikum Der Universität zu Köln, Cologne

IPD SHARING:
Plan to Share IPD: No
Participants have not provided informed consent for their anonymized individual data to be made available beyond that described in the patient information sheet.

REFERENCES:
- [Background] Asjo B, Stavang H, Sorensen B, Baksaas I, Nyhus J, Langeland N. Phase I trial of a therapeutic HIV type 1 vaccine, Vacc-4x, in HIV type 1-infected individuals with or without antiretroviral therapy. AIDS Res Hum Retroviruses. 2002 Dec 10;18(18):1357-65. doi: 10.1089/088922202320935438. PMID 12487807
- [Background] Kran AM, Sorensen B, Nyhus J, Sommerfelt MA, Baksaas I, Bruun JN, Kvale D. HLA- and dose-dependent immunogenicity of a peptide-based HIV-1 immunotherapy candidate (Vacc-4x). AIDS. 2004 Sep 24;18(14):1875-83. doi: 10.1097/00002030-200409240-00003. PMID 15353973
- [Background] Kvale D, Kran AM, Sommerfelt MA, Nyhus J, Baksaas I, Bruun JN, Sorensen B. Divergent in vitro and in vivo correlates of HIV-specific T-cell responses during onset of HIV viraemia. AIDS. 2005 Mar 24;19(6):563-7. doi: 10.1097/01.aids.0000163932.76531.c6. PMID 15802974
- [Background] Sommerfelt MA, Nyhus J, Sorensen B. Novel peptide-based HIV-1 immunotherapy. Expert Opin Biol Ther. 2004 Mar;4(3):349-61. doi: 10.1517/14712598.4.3.349. PMID 15006729

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Lenalidomide 5 mg: Intradermal Vacc-4x (1.2 mg) given with Leukine® (rhu-GM-CSF) (0.06 mg) and oral lenalidomide 5 mg
- Part A: Lenalidomide 10 mg: Intradermal Vacc-4x (1.2 mg) given with Leukine® (rhu-GM-CSF) (0.06 mg) and oral lenalidomide 10 mg
- Part A: Lenalidopmide 25 mg: Intradermal Vacc-4x (1.2 mg) given with Leukine® (rhu-GM-CSF) (0.06 mg) and oral lenalidomide 25 mg
Period: Overall Study
Arm/Group | Part A: Lenalidomide 5 mg | Part A: Lenalidomide 10 mg | Part A: Lenalidopmide 25 mg | Part B: Lenalidomide | Part B: Lenalidomide Placebo
Started | 3 | 3 | 6 | 12 | 12
Completed | 3 | 3 | 6 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Lenalidomide 5 mg | Part A: Lenalidomide 10 mg | Part A: Lenalidopmide 25 mg | Part B: Lenalidomide | Part B: Lenalidomide Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (4.16) | 35.7 (3.06) | 46.2 (5.42) | 44.4 (7.97) | 41.5 (8.04) | 42.9 (7.34)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 6 | 12 | 12 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 12 | 12 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1
  White | 3 | 1 | 6 | 12 | 11 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (2.32) | 27.9 (7.65) | 24.4 (1.75) | 23.6 (3.85) | 23.5 (3.44) | 24.1 (3.74)

OUTCOME MEASURES:

1. Primary Outcome: Part A: To Establish Highest Tolerated Dose of Lenalidomide, Dose-Limiting Toxicity
Description: Number of participants in each of the three groups that experienced any dose-limiting toxicity.
Time Frame: 31 days
Population: ITT analysis set was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Lenalidomide 5 mg | Part A: Lenalidomide 10 mg | Part A: Lenalidopmide 25 mg
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 0

2. Primary Outcome: Part A: To Establish Highest Tolerated Dose of Lenalidomide, CD4 Counts Over Time
Time Frame: 31 days
Population: ITT analysis set was used.
Measure: Mean (Standard Deviation); unit: 10^6 cells/mL
Arm/Group | Part A: Lenalidomide 5 mg | Part A: Lenalidomide 10 mg | Part A: Lenalidopmide 25 mg
Number analyzed (Participants) | 3 | 3 | 6
10^6 cells/mL
  Baseline | 437.3 (38.30) | 436.3 (60.05) | 454.2 (86.59)
  Week 1 | 393.0 (167.56) | 317.0 (18.52) | 342.2 (27.13)
  Week 4 | 442.0 (121.77) | 399.3 (15.95) | 450.7 (147.02)
  Week 5 | 432.7 (242.47) | 449.0 (71.04) | 452.3 (66.28)

3. Primary Outcome: Part B: Change in CD4 Count
Description: Change in CD4 count from baseline to Week 26.
Time Frame: Week 26
Population: Analysis was performed for both the Intent To Treat (ITT) and Per Protocol (PP) analysis set.
Measure: Mean (Standard Deviation); unit: 10^6 cells/L
Arm/Group | Part B: Lenalidomide | Part B: Lenalidomide Placebo
Number analyzed (Participants) | 12 | 12
10^6 cells/L
  ITT | 90.9 (98.79) | 42.2 (81.40)
  PP: number analyzed (Participants) | 10 | 11
  PP | 106.3 (101.00) | 49.1 (81.58)

4. Secondary Outcome: Part B: Change in CD8 Count
Description: Change in CD8 count from baseline to week 26.
Time Frame: 26 weeks
Population: Not all patients had quantifiable blood samples/counts at all time points
Measure: Mean (Standard Deviation); unit: 10^6 cells/L
Arm/Group | Part B: Lenalidomide | Part B: Lenalidomide Placebo
Number analyzed (Participants) | 12 | 12
10^6 cells/L
  Baseline | 734.2 (473.14) | 655.3 (325.19)
  Week 1: number analyzed (Participants) | 11 | 10
  Week 1 | 653.8 (382.16) | 784.5 (372.96)
  Week 4: number analyzed (Participants) | 12 | 11
  Week 4 | 744.9 (485.49) | 794.5 (452.91)
  Week 12 | 823.0 (548.84) | 760.3 (432.79)
  Week 13: number analyzed (Participants) | 12 | 11
  Week 13 | 811.2 (557.52) | 663.6 (393.95)

5. Secondary Outcome: Part B: Evaluate the Effect on HIV Viral Load
Description: Results BLQ (<20 HIV copies/mL) have been replaced with BLQ/2 = 10 HIV copies/mL while 'not detected' results have been replaced with 0 HIV copies/mL.
Time Frame: 26 weeks
Population: ITT analysis set
Measure: Mean (Standard Deviation); unit: Copies/mL
Arm/Group | Part B: Lenalidomide | Part B: Lenalidomide Placebo
Number analyzed (Participants) | 12 | 12
Copies/mL
  Baseline | 0.8 (2.89) | 2.5 (4.52)
  Week 1 | 5.1 (9.30) | 0.0 (0.00)
  Week 4: number analyzed (Participants) | 12 | 11
  Week 4 | 6.4 (8.17) | 0.9 (3.02)
  Week 12 | 5.5 (11.29) | 4.3 (6.90)
  Week 13 | 7.4 (19.77) | 1.7 (3.89)
  Week 21 | 1.7 (3.89) | 4.2 (5.15)
  Week 26 | 3.5 (6.99) | 2.5 (4.52)

6. Secondary Outcome: Part B: Incidents of Delayed-type Hypersensitivity
Description: Delayed-type hypersensitivity measured by induration and erythema.
Time Frame: 26 weeks
Population: The IIT population was used for this outcome measure. Data for one patient was not reported at week 26.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Lenalidomide | Part B: Lenalidomide Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Week 1, Induration | 0 | 0
  Week 1, Erythema | 0 | 1
  Week 26, Induration: number analyzed (Participants) | 11 | 11
  Week 26, Induration | 5 | 2
  Week 26, Erythema: number analyzed (Participants) | 11 | 11
  Week 26, Erythema | 6 | 6

7. Secondary Outcome: Part A and B: Safety and Tolerability
Time Frame: Part A: 31 days and Part B: 26 weeks
Measure: Number; unit: participants
Arm/Group | Part A: Lenalidomide 5 mg | Part A: Lenalidomide 10 mg | Part A: Lenalidopmide 25 mg | Part B: Lenalidomide | Part B: Lenalidomide Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 12 | 12
participants
  With any TEAE | 3 | 2 | 6 | 10 | 9
  With TESAE | 0 | 0 | 0 | 1 | 0
  With any AE resultiung in withdrawal | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing informed consent and until last visit; 31 days in Part A and 26 weeks in Part B. In addition, a 5-year survival follow-up period during which telephone contact from site for all subjects who discontinue treatment at any time will be conducted every 4 months for the first two years and every 6 months thereafter for a minimum of 5 years post-inclusion for survival, cause(s) of death, disease progression and post-treatment therapy(ies).
Arm/Group | Part A: Lenalidomide 5 mg | Part A: Lenalidomide 10 mg | Part A: Lenalidopmide 25 mg | Part B: Lenalidomide | Part B: Lenalidomide Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 6/6 | 10/12 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Lenalidomide 5 mg (N=3) | Part A: Lenalidomide 10 mg (N=3) | Part A: Lenalidopmide 25 mg (N=6) | Part B: Lenalidomide (N=12) | Part B: Lenalidomide Placebo (N=12)
Abscess left upper arm (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Lenalidomide 5 mg (N=3) | Part A: Lenalidomide 10 mg (N=3) | Part A: Lenalidopmide 25 mg (N=6) | Part B: Lenalidomide (N=12) | Part B: Lenalidomide Placebo (N=12)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (6)
Injection site erythema (General disorders) | 2 (4) | 1 (4) | 2 (2) | 4 (6) | 2 (3)
Injection site pruritus (General disorders) | 2 (4) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Injection site swelling (General disorders) | 1 (3) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Injection site warmth (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (6) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sunisitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (5) | 0 (0)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Abdominnal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Grand mal convultion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypogonadism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Listless (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor (or designee) will prepare a final report on the study. The Investigator may not publish or present any information on this study without the express written approval of the Sponsor. Additionally, the Sponsor, may, for any reason, withhold approval for publication or presentation.